CLINICAL TRIAL: NCT06598072
Title: Clinical Study to Evaluate the Efficacy of a Regimen Including Rinsing With an Alcohol Free Mouthwash Containing CPC+Zn as Compared to Dental Flossing and Brushing and a Regimen Including Rising With an Essential Oils Containing Alcohol Mouthwash in Reducing Dental Plaque and Gingivitis.
Brief Title: Comparative Study to Evaluate the Efficacy of an Alcohol-free Mouthwash Regimen With CPC+Zn, Flossing and Brushing, and an Alcohol-based Mouthwash Regimen With Essential Oils in Reducing Plaque and Gingivitis.
Acronym: PGMWII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Collaborators: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2024-08-PG-MWII-MX-CB
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-04-14 (Actual); Status verified 2025-04

CONDITIONS: Gingival Bleeding; Plaque Induced Gingival Disease; Gingival Diseases; Gingivitis and Periodontal Diseases
Keywords: gingivitis; dental plaque
MeSH Terms: conditions — Gingival Hemorrhage; Gingival Diseases; Gingivitis; Periodontal Diseases; Dental Plaque | interventions — Dental Devices, Home Care

STUDY DESIGN:
Intervention Model Description: This is a Phase III, randomized, controlled, double-blind, parallel-group clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking involves several key roles to ensure unbiased results and to maintain the integrity of the study results. The Participant, Care Provider, Investigator, and Outcomes Assessor are all masked in this double-blind study. The participants do not know which group they have been assigned to, the care providers administering the treatments are unaware of the specific products being used by each participant, the investigators conducting the study do not know the group assignments, and the outcomes assessors evaluating the results are blind to the treatment allocations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CPC+Zn mouthwash and brushing (Experimental): A regimen composing of a CPC+Zn mouthwash, brushing with a commercially available toothbrush and a stannous fluoride-based toothpaste
  Interventions: Drug: Mouthwash CPC+Zn+F
- Essential oils mouthwash and brushing (Active Comparator): A regimen composing of an essential oils mouthwash, brushing with a commercially available toothbrush and a fluoride-based toothpaste
  Interventions: Drug: Essential oils mouthwash
- Flossing and brushing (Active Comparator): A regimen composing of flossing and brushing with a commercially available toothbrush and a fluoride-based toothpaste
  Interventions: Device: Dental floss

INTERVENTIONS:
Drug: Mouthwash CPC+Zn+F — A mouthwash containing CPC + Zn and fluoride
  Other Names: CPC+Zn
  Arms: CPC+Zn mouthwash and brushing
Drug: Essential oils mouthwash — Essential oils mouthwash
  Arms: Essential oils mouthwash and brushing
Device: Dental floss — Dental Floss
  Arms: Flossing and brushing

SUMMARY:
This is a Phase III, randomized, one-center, parallel group, double blinded, clinical study to evaluate the efficacy of an alcohol-free mouthwash containing CPC+Zn as compared to dental flossing and to rising with an essential oils containing alcohol mouthwash in reducing dental plaque and gingivitis. One hundred and twenty participants, aged between 18 and 65 years, will be included and followed for 12 weeks.

DETAILED DESCRIPTION:
This clinical study aims to evaluate the efficacy of a regimen including an alcohol-free mouthwash containing CPC+Zn as compared to dental flossing and brushing and to a regimen including a rinsing with an essential oils containing alcohol mouthwash in reducing dental plaque and gingivitis. This is a Phase III, randomized, one-center, parallel group, double blinded, involving 120 participants, aged 18 to 65. Subjects will be allocated into 3 groups: one - using the CPC+Zn mouthwash, another using the essential oils mouthwash and a control group using dental floss. Each group will also use a fluoride toothpaste and a soft-bristle toothbrush twice daily over 12 weeks. The primary efficacy variable is the reduction of gingival inflammation also Probing Depth, Bleeding on Probing, and a Plaque Index will be accessed. Subjects will undergo baseline, 4-week, and 12-week evaluations, with data analyzed using ANCOVA to assess the efficacy and safety of the products. Adverse events and compliance will be closely monitored, with strict confidentiality maintained for all participants. The study rigorous design aims to provide comprehensive insights into the effectiveness of these oral hygiene regimens.

ELIGIBILITY:
Inclusion Criteria:

Availability for the duration of the study; Good general health (absence of any condition that, in the opinion of the Principal Investigator, might constitute a risk to the subject while participating in the study. Examples include heart problems, valve/hip replacements, etc); Willingness to provide information related to their medical history; At least 20 teeth with scorable facial and lingual surfaces; evidence of gingivitis; At least 10 bleeding sites based on the Bleeding Index (BI); Initial mean gingivitis index of at least 1.5 as determined by the use of the Modified Gingival Index (MGI); Subjects without allergies to the products that are being tested; Informed Consent Form signed.

Exclusion Criteria:

No sites with more than 5 mm probing depth, and a maximum of three sites of 5 mm probing depth.

Have received dental prophylaxis within 1 month prior to the Baseline visit; Need for antibiotics prior to dental treatment; use of antibiotics, anti-inflammatory or anticoagulant therapy during the three months prior to entry into the study; Usage of oral care products containing chemotherapeutic products within 2 weeks prior to Baseline; Use of smokeless tobacco; Any other condition that would make the volunteer inappropriate for the study. Oral pathology, chronic disease, or a history of allergy to testing products; Subject using anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti-inflammatory medication or daily analgesics within one month prior to the start of the study or scheduled to start such intake during the course of the study; Subject participating in any other clinical study; Subject pregnant or breastfeeding; Subject allergic to oral care products, personal care consumer products, or their ingredients; Ongoing use of medications known to affect the gingival tissues (i.e. calcium channel blockers, phenytoin, cyclosporine); Periodontal treatment 12 months before the beginning of the study; Current smokers and subjects with a history of alcohol or drug abuse; Subjects with orthodontic appliances or presence of fixed or removable prosthodontics dentures that may interfere with the evaluations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Modified Gingival Index | 12 weeks
  The Modified Gingival Index (MGI) is used to evaluate the severity of gingivitis by measuring the extent of gingival inflammation. It categorizes gingival health/inflammation on a scale from 0 to 4, where 0 signifies normal gingiva with no inflammation, and 4 indicates severe inflammation characterized by erythema, edema, and spontaneous bleeding.

SECONDARY OUTCOMES:
Turesky modification of Quigley-Hein Plaque Index | 12 weeks
  The Turesky modification of the Quigley-Hein Plaque Index is a method for assessing dental plaque accumulation by scoring plaque presence on six surfaces of each tooth on a scale from 0 to 5.
Bleeding on probing | 12 weeks
  Bleeding on probing (BOP) is a diagnostic technique used to assess gingival inflammation by gently probing the gum tissue; the presence of bleeding indicates inflammation and potential periodontal disease.
Probing depth | 12 weeks
  Probing depth measures the distance between the gingival margin and the bottom of the periodontal pocket using a calibrated periodontal probe, indicating the severity of periodontal disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Autónoma de San Luis Potosí, San Luis Potosí City, San Luis Potosí, Mexico

IPD SHARING:
Plan to Share IPD: No